CLINICAL TRIAL: NCT05600088
Title: Clinical Investigation of Intracoronary Cryotherapy Using the CryoTherapy System (CTS) for High-risk Plaque in Patients With (Non-)ST-segment Elevation Myocardial Infarction (NSTEMI) or Unstable Angina
Brief Title: Intracoronary Cryotherapy Effect on Stabilization of Vulnerable Plaque in Patients With (N)STEMI or Unstable Angina
Acronym: POLARSTAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cryotherapeutics SA (Industry)
Collaborators: CoreAalst BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CT-CD-P03-1
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease; Coronary Syndrome; Cryotherapy Effect; Myocardial Infarction; Myocardial Disease; Atherosclerosis, Coronary
MeSH Terms: conditions — Coronary Artery Disease; Angina, Unstable; Myocardial Infarction; Cardiomyopathies

STUDY DESIGN:
Intervention Model Description: up to 10 subjects with NSTEMI or unstable angina undergoing cryotherapy treatment of coronary vulnerable plaque lesions. Once This safety cohort has been enrolled, additional 20 subjects will be enrolled to further confirm feasibility and safety of the device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CTS Treatment Arm (Experimental): active cryotherapy of a single suitable high-risk coronary plaque lesion with CTS device
  Interventions: Device: CryoTherapy System (CTS)

INTERVENTIONS:
Device: CryoTherapy System (CTS) — local cryotherapy of coronary high-risk plaque lesions using the CTS consisting of a semi-compliant balloon and a console controlling the temperature of cryotherapy

SUMMARY:
The POLARSTAR study is an early safety and feasibility study to evaluate the performance and safety of the CryoTherapy System (CTS) for the treatment of coronary plaque lesions that are not obstructing blood flow but are at high-risk of rupture which would cause a major heart attack. The CTS is used to apply local freezing of the lesion using a balloon catheter, controlled by a console that regulates in- and outflow of a cooling agent into the catheter. The treatment is expected to stabilize the lesion, diminishing the risk of rupture. The study will enrol subjects with acute coronary disease who have suitable coronary lesions. Subjects will be followed for 1 year after the CTS treatment. Baseline identification of lesions will be done using Coronary CT-angiography (CCTA), which will be repeated at 3 and 9 months after procedure.

DETAILED DESCRIPTION:
The POLARSTAR study is an early feasibility study to evaluate the safety and performance of the CryoTherapy System (CTS) medical device, consisting of a console and a balloon catheter. The CTS is designed to deliver local cryo-energy to vulnerable plaque lesions in the coronary arteries, aiming to stabilize the plaque to reduce the risk of rupture and subsequent cardiac events. The study will enrol up to 10 subjects with NSTEMI or unstable angina, who underwent successful Percutaneous Coronary Intervention (PCI) of their culprit coronary lesion, and who were identified to have presence of at least 1 non-culprit suitable plaque lesion at high-risk of rupture. After providing informed consent the subjects will undergo a Coronary CT-angiography (CCTA) to confirm suitability of the coronary plaque lesion. A single high-risk plaque lesion will be treated by the investigators, with Intra-vascular Ultrasound (IVUS) imaging prior to and after CTS treatment. Subjects will be followed clinically for up to one year after the CTS treatment, and will have follow-up CCTA assessments at 3 and 9 months post-procedure. Primary endpoint will be Major cardiac events rate at 3 months post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old.
2. Subject has acute cardiac pain/angina consistent with acute coronary syndrome eligible for coronary angiography meeting one of the following criteria:

   1. (Non-)ST-segment elevation myocardial infarction ((N)STEMI) with rise/fall of cardiac enzymes (troponin I or T) with at least one value above the 99th percentile of the upper reference limit requiring PCI within 72 hours from diagnosis
   2. Unstable angina
3. Successful PCI (defined as diameter stenosis less than 30% and TIMI 3 flow on final angiography without procedural complication) of the culprit lesion.
4. Subject has at least one high-risk plaque meeting the criteria below:

   1. Located in a non-culprit vessel,
   2. High-risk plaque lesion on CCTA and at least one of the following features:

      1. Presence of low-attenuation plaque (HU<50) and/or
      2. Positive remodelling (remodelling index >1.1) and/or
      3. Napkin ring sign and/or
      4. Plaque burden ≥70%
   3. Lesion length ≤ 20 mm.
   4. Diameter stenosis on invasive angiography between 30% and 70% on coronary angiogram or negative physiology assessment (FFR>0.80 or non-hyperemic pressure ratios (NHPR) >0.89).
   5. Reference vessel diameter (RVD) < 3.75 mm and > 2.00 mm in diameter
   6. Investigator considers that lesions are accessible.
   7. If more than two suitable lesions available, investigator will select the most appropriate lesion for cryotherapy treatment.
5. Subject is able to provide consent and has signed and dated the informed consent form.

Exclusion Criteria:

1. Subject is hemodynamically unstable (cardiogenic shock, hypotension needing inotropes, hypoxia needing intubation, refractory ventricular arrhythmias, and IABP).
2. Subject has ongoing ST-segment elevation myocardial infarction.
3. Subject had a procedural complication during the Acute coronary syndrome (ACS) PCI procedure.
4. Subject has history of Coronary Artery Bypass Graft (CABG) or planned CABG within 12 months after the index procedure.
5. Subject has known reduced Left Ventricular Ejection Fraction < 30%.
6. Subject has known severe valvular heart disease.
7. Subject has known severe renal insufficiency (eGFR <30 ml/min/1.72 m2).
8. Subject has any life-threatening conditions or medical comorbidity resulting in life expectancy < 12 months.
9. Subject is currently participating in another clinical investigation that has not yet reached its primary endpoint.
10. Subject is pregnant or lactating, or NOT surgically sterile (tubal ligation or hysterectomy) or NOT postmenopausal for at least 6 months or is a female with childbearing potential without effective contraception (pill, patch, ring, diaphragm, implant and intrauterine device).

Angiographic exclusion criteria:

1. Visible distal embolization/no-reflow following culprit lesions PCI.
2. Left main coronary artery disease (visual diameter stenosis > 50%).
3. Stent thrombosis/restenosis as a culprit lesion.
4. CTS lesion involving a bifurcation (defined as lesions involving side branches >2.0 mm).
5. Angiographic or CCTA evidence of severe calcification and/or marked tortuosity of the index vessel and/or lesion.
6. Thrombotic lesions
7. Ostial lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety: Rate of Cryotherapy related adverse events | 90 days post-procedure
  Any cryotherapy procedure related complication defined as coronary artery dissection (angiographic dissection ≥ NHLBI type B), acute vessel closure, life threatening arrythmia, need for bailout stenting, or any Major Adverse Cardia Event (MACE) defined as cardiac death, CTS-treated vessel myocardial infarction, CTS-treated lesion revascularization, rehospitalization for unstable or progressive angina adjudicated to the CTS-treated lesion

SECONDARY OUTCOMES:
Safety: Rate of Cryotherapy related events | 1 year post-procedure
  Any cryotherapy procedure related complication defined as coronary artery dissection (angiographic dissection ≥ NHLBI type B), acute vessel closure, life threatening arrythmia, need for bailout stenting, or any MACE defined as cardiac death, CTS-treated vessel myocardial infarction, CTS-treated lesion revascularization, rehospitalization for unstable or progressive angina adjudicated to the CTS-treated lesion
Device success | end of CTS treatment
  Number of lesions successfully treated without device deficiency
CTS procedure success | end of CTS treatment
  Number of lesions successfully treated to obtain Thrombolysis in Myocardial Infarction (TIMI) 3 flow
Imaging: CCTA assessed Minimum lumen area (MLA) | 90 days post-procedure
  Change in MLA (mm²) compared to baseline
Imaging: CCTA assessed Minimum lumen area (MLA) | 9 months post-procedure
  Change in MLA (mm²) compared to baseline
Imaging: CCTA assessed area stenosis | 3 months post-procedure
  Change in area stenosis % compared to baseline
Imaging: CCTA assessed area stenosis | 9 months post-procedure
  Change in area stenosis % compared to baseline
Imaging: CCTA assessed lesion plaque burden | 3 months post-procedure
  Change in lesion plaque burden % from baseline
Imaging: CCTA assessed lesion plaque burden | 9 months post-procedure
  Change in lesion plaque burden from baseline
Imaging: CCTA assessed Total plaque volume | 3 months post-procedure
  Change in total plaque volume (mm³) from baseline
Imaging: CCTA assessed Total plaque volume | 9 months post-procedure
  Change in total plaque volume(mm³) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Irakli Gogorishvili, MD, Principal Investigator — Israeli_Georgian research Clinic Helsicore, Tbilisi, Georgia
Locations (5):
- Georgia (2):
  - Israeli-Georgian Research Clinic Helsicore, Tbilisi
  - Tbilisi Heart Center, Tbilisi
- Lithuania (3):
  - Hospital of Lithuanian University of health sciences Kauno Klinikos, Kaunas
  - Klaipèda University Hospital, Klaipèda
  - Vilnius University Hospital Santaros Klinikos, Vilnius

IPD SHARING:
Plan to Share IPD: No